CLINICAL TRIAL: NCT03377517
Title: A Pilot Study of Stereotactic Radiosurgical Hypophysectomy for Intractable Pain From Bone Metastases
Brief Title: Radiosurgical Hypophysectomy for Bone Metasteses Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual was slower than anticipated and funding was not extended beyond original contract.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Accuray Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J17181; IRB00158648 (Other: JHM IRB)
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Bone Metastases

STUDY DESIGN:
Intervention Model Description: Patients will be treated to a dose of 150 Gy in a single fraction. All patients will undergo CT simulation with 1 mm slices as well as MRI simulation including at least high resolution 1 mm slice T1 weighted MRI. They will be treated in a supine position using an aquaplast mask system for immobilization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ResearchTreatment Plan (Experimental): Patients will be treated to a dose of 150 Gy in a single fraction. All patients will undergo CT simulation with 1 mm slices as well as MRI simulation including at least high resolution 1 mm slice T1 weighted MRI. They will be treated in a supine position using an aquaplast mask system for immobilization.
  Interventions: Radiation: radiosurgical hypophysectomy

INTERVENTIONS:
Radiation: radiosurgical hypophysectomy — Patients will be treated to a dose of 150 Gy in a single fraction. All patients will undergo CT simulation with 1 mm slices as well as MRI simulation including at least high resolution 1 mm slice T1 weighted MRI. They will be treated in a supine position using an aquaplast mask system for immobilization.

SUMMARY:
This research is being done to see if a delivery of a single high dose of radiation therapy to a small area of the pituitary gland and pituitary stalk in a highly precise manner may be helpful in reducing intractable pain from bone metastases.

DETAILED DESCRIPTION:
Although not currently standard of care, small series suggest both safety and efficacy of radiosurgical hypophysectomy in reducing cancer pain from bone metastases. In spite of the demonstrated feasibility in meeting normal tissue constraints and preliminary data suggestive of both safety and efficacy, radiosurgical hypophysectomy is rarely performed in clinical practice, and many radiation oncologists are not even aware of its potential to reduce intractable cancer pain. This is likely because, to date, well-designed prospective studies have not been performed to further explore both the safety and efficacy of the intervention. This single arm pilot study is designed to fill that void. If successful, the investigators plan to utilize the data to support the proposal of a larger scale follow-up clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologic proof of malignancy
2. Radiographic evidence of bone metastases
3. Intractable pain uncontrolled by opioids, medical management, injections/ablation or surgical intervention that would be difficult to address with conventional radiation therapy or other standard options and is limiting the patient's function and quality of life. Intractable pain will be defined as a visual analogue score of at least 4.
4. Definitive radiographic progression of osseous and/or visceral metastases on standard staging scans (CT, MRI, bone scan, PET scan or any other standard of care imaging) performed within the last 3 months in spite of standard oncologic interventions and/or inability to tolerate standard oncologic interventions
5. Life expectancy at least 4 weeks
6. Age≥ 18 years
7. Patients of childbearing potential (male or female) must practice adequate contraception due to possible harmful effects of radiation therapy on an unborn child
8. Patient must have the ability to understand and the willingness to sign a written informed consent document
9. All patients must be informed of the investigational nature of this study and must be given written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

1. Prior brain radiation
2. Patients must not have a serious medical or psychiatric illness that would, in the opinion of the treating physician prevent informed consent or completion of protocol treatment
3. Isolated localized pain amenable to focal radiation therapy, or pain well controlled by opioids, medical management, injections/ablation or surgical intervention
4. Malignancies being managed with curative intent
5. Life expectancy <4 weeks
6. The tumor amenable to curative management

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Intensity of Bone Pain | 4 weeks
  To estimate the rate of clinically meaningful decrease in diffuse osseous pain following radiosurgical hypophysectomy at 4 weeks following completion of radiosurgical hypophysectomy

SECONDARY OUTCOMES:
Rate of change of disease spread | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the rate of clinically meaningful decrease in diffuse osseous pain following radiosurgical hypophysectomy
Rate of Change of Quality of Life | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the rate of clinically meaningful increase in patient reported quality of life following radiosurgical hypophysectomy
Rate of change in opioid use | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the rate of reduction in opioid utilization following radiosurgical hypophysectomy
Rate of biochemical endocrinopathy | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the rate of biochemical endocrinopathy following radiosurgical hypophysectomy
Rate of change of optic nueropathy | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the risk of radiation induced optic neuropathy following radiosurgical hypophysectomy
Rate of change of neurologic toxicity | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the radiation-associated acute and long term neurologic toxicity of radiosurgical hypophysectomy
Rate of change of insipidus diabetes | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the rate of diabetes insipidus following radiosurgical hypophysectomy
Rate of change in costs | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the cost effectiveness of radiosurgical hypophysectomy
Rate of change of cortisol | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the relationship between pain response and cortisol levels
Rate of change of pain with respect to hormones | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the rate of pain response in hormonally active and non-hormonally active tumors
Rate of change of pain with respect to morphine | Up to 100 weeks following completion of radiosurgical hypophysectomy
  To estimate the rate of pain response in morphine sensitive and morphine insensitive tumors

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Redmond, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehsensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No